CLINICAL TRIAL: NCT02074137
Title: Multicentre, Single Arm, Open Label, Non Controlled Phase IV Clinical Trial to Evaluate Safety of Cabazitaxel (Jevtana) in Combination With Oral Prednisone (or Prednisolone) for the Treatment of Patients With Metastatic Hormone Refractory Prostate Cancer Previously Treated With a Docetaxel-containing Regimen
Brief Title: Evaluation of Safety of Cabazitaxel (Jevtana) in Patients With Metastatic Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABAZL06499; U1111-1131-3161 (Other: UTN)
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Last update posted 2016-06-02 (Estimated); Status verified 2016-06

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabazitaxel (Experimental): Cabazitaxel 25 mg/m² intravenously every 3 weeks, in combination with oral prednisone or prednisolone 10 mg daily
  Interventions: Drug: CABAZITAXEL XRP6258; Drug: Prednisone; Drug: Prednisolone

INTERVENTIONS:
Drug: CABAZITAXEL XRP6258 — Pharmaceutical form:Solution Route of administration: Intravenous
Drug: Prednisone — Pharmaceutical form:Tablet Route of administration: Oral
Drug: Prednisolone — Pharmaceutical form:Tablet Route of administration: Oral

SUMMARY:
Primary Objective:

To evaluate the safety of cabazitaxel (Jevtana) in patients with metastatic hormone refractory prostate cancer

Secondary Objectives:

1. To describe the use of cabazitaxel (Jevtana) in combination with oral prednisolone for the treatment of patients with metastatic Hormone Refractory Prostate Cancer
2. To describe patient profile in terms of demography, disease characteristics and prior treatment history
3. To describe efficacy outcomes: radiological response (if available) using Recist criteria V 1.1 and Prostate Specific Antigen (PSA) response

DETAILED DESCRIPTION:
The study consists of:

* a screening phase (maximum length of 7-day).
* a treatment phase with 21-day study treatment cycles. Patients continue to receive treatment until disease progression , death, unacceptable toxicity, investigator's decision or withdrawal of consent.
* a 30-day follow-up visit after the last dose of study medication.

ELIGIBILITY:
Inclusion criteria :

* Metastatic hormone refractory prostate cancer (mHRPC) previously treated with a docetaxel-containing regimen
* Disease Progression during or after docetaxel-containing regimen for mHRPC
* Surgical or medical castration
* Patient is ≥ 18 years and ≤ 75 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Adequate bone marrow, liver, and renal function: Neutrophils> 1500 /mm3; Hemoglobin > 10 g/dL; Platelets > 100 x109/L; Bilirubin < Upper Normal Limit (ULN); Serum Glutamate Oxaloacetate Transaminase (Aspartate Aminotransferase)/SGOT (AST) < 1.5xULN; Serum Glutamate Pyruvate Transaminase (Alanine Aminotransferase)/SGPT (ALT) < 1.5xULN; Creatinine < 1.5xULN. In case of creatinine > 1.0 x ULN and < or = 1.5 x ULN, calculated creatinine clearance according to CKD-EPI formula should be > or = 60 ml/min.
* Written informed consent must be obtained prior to any study related procedures

Exclusion criteria:

* Prior radiotherapy to ≥ 40% of bone marrow
* Previous treatment with cabazitaxel (Jevtana®)
* Prior surgery, radiation, chemotherapy, or other anti-cancer therapy within 4 weeks prior to enrollment
* Active grade ≥2 peripheral neuropathy
* Active grade ≥2 stomatitis
* Active infection requiring systemic antibiotic or anti-fungal medication
* Active cancer (other than mHRPC) including prior malignancy from which the patient has been disease-free for ≤5 years
* Known brain or leptomeningeal involvement
* History of severe hypersensitivity reaction (≥grade 3) to docetaxel
* History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs
* History of severe hypersensitivity reaction (≥grade 3) or intolerance to prednisone or prednisolone
* Uncontrolled severe illness or medical condition (including uncontrolled diabetes mellitus)
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (a 2 weeks wash-out period is necessary for patients who are already on these treatments). Participation in any other clinical trial with any investigational drug
* Patient with reproductive potential not implementing accepted and effective method of contraception

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with Related Serious Adverse Events | up to13 months

SECONDARY OUTCOMES:
Evaluation of use of cabazitaxel in terms of treatment duration, number of cycles, dose modifications | up to 13 months
Radiological overall response (if radiological tumor assessment done) using Recist criteria | up to 13 months
Number of patients with at least 50% decrease in PSA | up to 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- India (3):
  - Investigational Site Number 356005, Kollkata
  - Investigational Site Number 356003, New Delhi
  - Investigational Site Number 356002, Trivandrum